CLINICAL TRIAL: NCT01553487
Title: Effects Of Unilateral Forearm Vibration On The Loss Of Muscle Strength And Bone Of The Contralateral Forearm Due to Forearm/Elbow Fracture
Brief Title: Effects Of Unilateral Forearm Vibration On The Loss Of Muscle And Bone Of Contralateral Forearm
Acronym: Vib-Frx
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not found voluntary subjects
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan Karacan, Clinical Associated Professor, Clinical Associated Professor, Bagcilar Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BEAH FTR-6
Record Dates: First submitted 2012-03-05; First posted 2012-03-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Effects of Vibration
Keywords: vibration; muscle strength; bone loss; immobilization; fracture
MeSH Terms: conditions — Bone Diseases, Metabolic; Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Excercise (Experimental): The forearm vibration training
  Interventions: Other: Forearm vibration
- Control (No Intervention): Patients will be treated by routine fracture treatment methods (fixation and rest).

INTERVENTIONS:
Other: Forearm vibration — All cases will be trained by forearm vibration device 5 times a week for six weeks period.
  Other Names: vibration training
  Arms: Excercise

SUMMARY:
The aim of the present study is to investigate the effects of vibrating the forearm bone in the free limb on muscle strength and bone mineral density of the forearm in patients with forearm/elbow fracture.

A total of 80 patients with forearm/elbow fracture are planned to include in this study. Patients will be randomly attained Training or Control group. Training period will be six weeks. Patients in the control group will receive standard care for provided for fractures, including fixation and rest.Before the start of the study and after six weeks, bilateral bone density of distal radius will be measured by DXA. Before trials, grip strength and the rest muscle electrical activity of contralateral wrist flexors and extensors will be measured. After six weeks, bilateral grip strength and the rest muscle electrical activity will be measured.

DETAILED DESCRIPTION:
The structure of a bone and the muscles surrounding it changes in a temporally synchronized fashion. Skeletal muscles have positive effects on bone structure and function. It is well-known that exercise training of muscles improves the resistance of bone to mechanical loading and that physical activity is also important for treating and preventing osteoporosis. Resistance and impact training can induce bone formation and/or prevent bone resorption. Immobilization frequently leads disuse osteoporosis in patients with a bone fracture.

Vibration has a strong osteogenic effect. The cyclic mechanical loading to the bone stimulates osteocytes. Vibration-induced bone formation is neuronally regulated. Vibration can also effectively enhance muscle strength and power. Previous studies have shown that vibration increases muscle electromyographic (EMG) activity. Based on the bone myoregulation reflex, bone is sensitive to mechanical stimuli and can send mechanical input signals to central nervous system and so can neuronally regulate the muscle activity.

Previous studies have documented the impact of unilateral training of limb muscle on the untrained contralateral homologous muscle.

The aim of the present study is to investigate the effects of vibrating the forearm bone in the free limb on muscle strength and bone mineral density of the forearm in patients with forearm/elbow fracture.

The study will include a total of 80 patients with forearm/elbow fractures. The participants meeting inclusion criteria will be randomized into one of two groups: a training group (40 cases) and a control group (40 cases). Patients in the control group will receive standard care for provided for fractures, including fixation and rest.

Forearm Vibration: Training group will exercise 5 times a week for six week period using a forearm vibration device. The forearm vibration device consists of a joystick unit, a weight-pulley system and a control panel. The subject will be seated in a chair. The right forearm will be placed on the vibration device with the shoulder in 10 degrees abduction, the elbow in 90 degrees flexion and the forearm and wrist in the neutral position. The axis of rotation of joystick unit will be aligned with that of the wrist joint of the free arm. The joystick unit will be capable of performing both an angular and a sliding motion simultaneously. The angular motion obtained the vibration effect and the sliding motion obtained the compression effect. The angular motion of the joystick unit will be provided by an electric motor. The range of angular motion will be 6 degrees. The weight is attached to the joystick with a rope and pulley system to provide mechanical loading to the forearm (compression effect). This weight is defined as vibration load. Maximum vibration load tolerated will be applied during vibration. The amplitude of vibration (range of motion of the wrist) will be 6 degree and the frequency of the vibration will be 40 Hz. The exercise duration and intensity will be low at the beginning but increased systematically over the 6-week training period. The subjects will be asked to report negative side effects or adverse reactions in their training diary.

Bone Densitometry: Before trails and after six weeks, bilateral bone density of distal radius will be measured by DXA. The bilateral bone density will be evaluated by bone densitometer (Norland).

Grip Strength Measurement: Before the start of the study, grip strength of wrist muscles in the free limb will be measured. After six weeks, bilateral grip strength will be measured by a hand dynamometer (Jamar digital plus hand dynamometer).

Surface EMG: Surface EMG of the right and left wrist muscles will be recorded using disposable self-adhesive bipolar Ag/AgCl electrodes (Kendall Arbo ) placed on its belly. The small disc electrodes (10-mm in diameter, inter-electrode distance of 20 mm) arranged in the direction of the muscle fibers. All cables will be carefully taped to the skin.

The skin overlying the muscle will be shaved, light abrasion will be applied, the skin will be cleaned using 70% alcohol and, conductive paste will be used to reduce electrode resistance before placing the electrodes.

Motor unit potentials will be amplified and recorded on a computer for off-line analyses at a sampling frequency of 2k using a data acquisition and analysis system (Powerlab data acquisition system, ADInstruments, Australia).

Twenty seconds of myoelectrical activity will be recorded from wrist muscles at rest. The mean myoelectrical activity will be calculated as the root mean squared (RMS) using the EMG device software, and defined as the "resting myoelectrical activity". The resting myoelectrical activity will be expressed as microvolt.

Power spectral analyses will be done. They will be conducted using Hamming windowed, 2048 point epochs, resulting in a frequency resolution of 0.98 Hz.

This is a prospective, randomized, controlled, single blind trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with a simple (uncomplicated) forearm/elbow fracture
* Males and females between 18 and 50 years of age

Exclusion Criteria:

* Fracture of distal radius
* Multiple previous fractures of bones in the upper extremities
* Complicated fracture (associated skin and/or tendon and/or nerve and/or vascular trauma, fragmented fractures )
* Patients not examined within the first three days after a trauma
* Upper extremity problems

  * Orthopedic problems: shortness of arms, congenital abnormalities
  * Joint disease (arthritis, joint prosthesis, etc.)
  * Other painful pathologies in the upper extremities (tendinitis, bursitis, etc.)
  * Circulation problems in the upper extremities
  * Skin lesions, dermatologic disorders
* Hypertension (>135 mmHg systolic, >85 mmHg diastolic) or Heart disease (coronary dis, conduction/rhythm prob, cardiac pacemaker)
* Neurological diseases (CNS problems, peripheral neuropathy)
* Systemic disease affecting bone metabolism: secondary osteoporosis, osteomalacia, Paget's disease, Diabetes mellitus, hepatic disease, renal dis. etc
* Non-cooperative patients, psychiatric conditions (panic attacks etc)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change of forearm muscle strength | baseline and 6 weeks
  Change of muscle strength with forearm vibration

SECONDARY OUTCOMES:
Change of distal radius bone mineral density | baseline and 6 weeks
  Change of distal radius bone mineral density with forearm vibration

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Study Chair — Bagcilar Training & Research Hospital
Locations (1):
- Bagcilar Training & Research Hospital, Istanbul, Turkey (Türkiye)